CLINICAL TRIAL: NCT00591669
Title: Non-invasive Imaging of GI Inflammation Using Microbubble Contrast Enhanced Ultrasonography
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data storage damage plus unexpected loss of funding
Sponsor: University of Virginia (Other)
Responsible Party: Brian Behm, MD, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 11971
Record Dates: First submitted 2007-12-26; First posted 2008-01-11 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory bowel disease; Crohn's disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease | interventions — perflutren

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IBD patients
  Interventions: Other: Definity
- 2 (Other): Control subjects
  Interventions: Other: Definity

INTERVENTIONS:
Other: Definity — We will be placing one vial (1.3) of Definity® in 50 mL of preservative-free saline. Our infusions will be initiated at slightly lower than recommended starting rate (3mL/min) and will be adjusted as necessary to produce optimal enhancement. The rate will not exceed 10 ml/min and we will not give more than 1.3 mL of Definity® in 50mL saline in any 24-hour period.
  Arms: 1
Other: Definity — We will be placing one vial (1.3) of Definity® in 50 mL of preservative-free saline. Our infusions will be initiated at slightly lower than recommended starting rate (3mL/min) and will be adjusted as necessary to produce optimal enhancement. The rate will not exceed 10 ml/min and we will not give more than 1.3 mL of Definity® in 50mL saline in any 24-hour period.
  Arms: 2

SUMMARY:
Inflammatory bowel disease (IBD) is a common chronic inflammatory disorder, but a noninvasive method of assessing disease location, severity, and extent is currently not available. Recently published animal data suggests that using transabdominal ultrasound enhanced with encapsulated gaseous microbubbles may provide a reliable, noninvasive means to detect and quantify areas of intestinal inflammation. This study will evaluate the role of Contrast-enhanced ultrasonography (CEU) for use as a diagnostic tool in patients with IBD. We hypothesize that the severity and extent of chronic intestinal inflammation, as quantified by CEU-derived video intensity scores, will correlate with endoscopically-derived measures of intestinal inflammation as obtained from the Crohn's Disease Endoscopic Inflammatory Index (CDEIS). A total of 40 patients will be enrolled in the study, 30 patients with IBD and 10 patients undergoing colonoscopy for other reasons. Prior to colonoscopy CEU assessment of small and large intestine will be performed to evaluate neoangiogenesis and intestinal blood flow. The correlation between the CEU-derived video intensity score and CDEIS will be assessed using Pearson's correlation coefficient. Subjects may also undergo scoring using the Rutgeerts Score, an endoscopic disease assessment index used to score disease activity in patients with previous ileocolonic resection. Comparing video intensity between IBD and non-IBD subjects will be performed using the Wilcoxon rank sum test, with a secondary aim of establishing preliminary estimates of the sensitivity of the microbubble scoring system.

DETAILED DESCRIPTION:
GI inflammation may indicate a number of complications or diseases, one of which is inflammatory bowel disease (IBD), now the second most prevalent inflammatory disorder in the world. Symptoms of the disease include severe abdominal pain, bloody diarrhea, persistent fever, weight loss, and significant malnutrition. There is also an increased risk of colon cancer. If left untreated, the disease is debilitating. Prompt intervention may reduce the amount of immunosuppressive therapy that is required to control the disease, but by the time the patient becomes symptomatic, the inflammatory response is difficult to suppress and much of the damage has already been done. It is therefore important to closely monitor patients with IBD. The location, extent, and severity of the inflammation are of primary consideration for correct diagnosis and treatment. However, no inexpensive and non-invasive procedure exists in protocol for the assessment of these factors of IBD. A non-invasive diagnostic that can detect the onset of inflammation and measure the extent of inflammatory involvement would be a valuable tool for the evaluation of patients with IBD.

Endoscopy, barium contrast X-ray studies, computed tomography (CT), magnetic resonance imaging (MRI), and transabdominal ultrasound (US) are currently the most common procedures used by gastroenterologists. The preferred manner of investigating GI inflammation includes endoscopy with biopsy, as only endoscopy can confirm the presence of inflammation. However, this procedure is highly invasive and limited to areas accessible to the endoscope. There are also limited but real risks associated with endoscopy. In addition, the cost of such a procedure may be prohibitive, or a qualified professional inaccessible, for some patients. Barium contrast X-ray studies remain the best way to visualize stricture and fistulae in the small intestine, but do not provide insight into the degree and extent of active inflammation. Repeated X-rays in chronic and younger patients also contribute to risk of irradiation. CT and MRI are the gold-standard for imaging extra-intestinal inflammatory disease, but fail in their ability to identify active inflammation. There have recently been many studies attempting to improve these means of assessing GI inflammation.

Transabdominal US presents a non-invasive means of imaging internal organs that imposes no significant health risks or undue discomfort upon the patient. The use of abdominal US for the evaluation of IBD was implemented as early as 1979, where wall thickening of the terminal ileum and cecum, with accompanying inflammatory changes in the mesentery, yielded recognizable patterns in both longitudinal and transverse images.11 These initial ultrasonographic images lacked sufficient resolution to provide a sensitive measure of disease activity, but technological advances in high frequency US have greatly improved resolution over the past twenty years. Still, the location and chronicity of certain conditions may decrease the efficacy of this imaging technique, making endoscopy the preferred method of investigation of GI problems. At present, there are several research groups actively investigating the application of US for the management of IBD. The combined results of these studies, in addition to the relatively wide availability, low cost, and easy use of US equipment, support the rationale for developing US into a useful tool for the evaluation of IBD.

Contrast-enhanced ultrasonography (CEU) is the main strategy for improving US quality. One contrast agent that has been studied in the imaging of inflammation, but which has not yet been human-tested for improvement of US quality in inflammation due to IBD, is microbubbles (MB). MB contrast agents are FDA-approved, and are becoming a common clinical tool for the enhancement of US imaging of cardiovascular hemodynamics around the world. Unlike tissue signal, which is produced by US reflection, the strong signal generated by MB is produced by radial oscillation of the MB in the acoustic field. Current MB used for perfusion imaging have lipid or albumin shells and contain high-molecular weight gases (perfluorocarbons, sulfur hexafluoride), which contribute to their high intravascular stability by preventing outward diffusion of gas. MB are generally 2-4µm in size - smaller than average capillary dimension - and passes unimpeded through the microcirculation. They are also hemodynamically inert, and behave similar to red blood cells in vivo. In animal models the acoustic properties of activated Definity® (Perflutren Lipid Microsphere) injectable suspension, were established at or below a mechanical index of 0.7 (1.8 MHz frequency). In clinical trials, the majority of the patients were imaged at or below a mechanical index of .08.

There are two ways that microbubbles might contribute to a strong signal in areas of inflammation in the small intestine or colon. The first is directly through neoangiogenesis and the increase in blood flow to the site. Defined as the growth of new blood vessels, neoangiogenesis is important to the pathogenesis of both Crohn's disease and ulcerative colitis. An expanded microvascular bed in the mucosa and submucosa of IBD patients with active inflammation has been confirmed, and is consistent with the high levels of integrins characteristic for proliferating endothelium (e.g. IL-8, bFGF, and VEGF) found in the microvessels of tissue affected by IBD. The hope is that the increased blood flow in actively inflamed IBD will be correlated with a stronger US signal from the increased concentration of MB flowing through the site.

The second way microbubble CEU may be effective at identifying active inflammation is an indirect effect of new microvasculature. Neoangiogenesis is thought to contribute to pathogenesis by fostering the recruitment and activation of an increased number of leukocyte into the inflamed mucosa. It has been observed that both albumin and lipid shell MB used for echocardiographic studies are phagocytosed intact by activated leukocytes, some of which are adherent to the inflamed endothelium of small intestine or colon. These phagocytosed MB retain a percentage of their acoustic properties, enabling US to image inflammation non-invasively in an in vivo setting. Incorporation of specific lipid moieties into the microbubble shell increases retention and phagocytosis by activated leukocytes.

An investigation of the efficacy of microbubble contrast agents in imaging GI inflammation is the first step towards such targeted imaging and tissue-targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inflammatory bowel disease (IBD), scheduled for diagnostic colonoscopy or
* Patients scheduled for diagnostic colonoscopy for other indications other than IBD (e.g. screening, family history of colon cancer).

Exclusion Criteria:

* Ineligibility for colonoscopy
* For control patients: a personal history of IBD or clinical history suspicious for IBD or other disease associated with intestinal inflammation. To be determined by investigators at the time of screening.
* Abnormal QT, Tic, or PR intervals during screening ECG
* Life-threatening ventricular arrhythmias during screening ECG
* Abnormally low oxygen saturation (<80%)
* History of the following:
* An intracardial or intrapulmonary shunt
* Unstable coronary artery disease
* Cerebrovascular disease (e.g. stroke or aneurysm)
* Diagnosed and or current signs or symptoms of severe, progressive or uncontrolled congenital heart failure
* Diagnosed and/or current signs or symptoms of severe, progressive or uncontrolled emphysema/COPD
* Diagnosed and/or current signs or symptoms of severe, progressive or uncontrolled pulmonary hypertension (known PA pressures >50mmHg)
* Uncontrolled high blood pressure (>140/90)
* Abnormal kidney function (creatinine > 2.0 mg/dl or GFR > 90)
* Abnormal liver function (Aspartate transaminase (AST), alanine transaminase (ALT), and alkaline phosphatase levels greater than 2 times the upper limit of normal.)
* Known hypersensitivity to octafluoropropane
* Pregnancy or nursing, confirmed by urine pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary study endpoint is to assess the degree of correlation of the video intensity score from microbubble imaging with an endoscopic scoring system for IBD, the Crohn's Disease Endoscopic Inflammatory Index (CDEIS). | Following data collection

SECONDARY OUTCOMES:
Secondary endpoint includes comparing the level of video intensity between 30 subjects with inflammatory bowel disease with 10 control patients who are undergoing endoscopic evaluation for non-inflammatory conditions of the large bowel. | Following data collection

CONTACTS AND LOCATIONS:
Overall Officials: Brian Behm, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States